CLINICAL TRIAL: NCT00182338
Title: Evaluation of Volume Status in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Scott Brimble, McMaster University
Other Study IDs: PD 04-2305
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Diseases; Inflammation; Peritoneal Dialysis
Keywords: cardiovascular outcomes; congestive heart failure; Peritoneal Membrane transport properties; Arterial stiffening; Inflammatory markers
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peritoneal Dialysis Patients

SUMMARY:
Patients with kidney failure on dialysis have a much higher risk of developing cardiovascular disease as compared to the general population. Recently, two large studies have shown that increasing the amount of dialysis does not decrease cardiovascular disease. It is known that retaining too much fluid leads to high blood pressure and thickening of the heart wall. Peritoneal dialysis is a method of home dialysis which allows dialysis patients autonomy and independence. This study will measure blood levels of a protein called N-BNP and measure the extent of body fluid by a machine called a bioimpedance analyzer. This device administers an undetectible electric current which distributes throughout total body water. The relationship between these tests and the clinical presence of volume expansion will be assessed. In addition, the extent of total body fluid and it's impact on heart attacks, heart failure and stroke will be determined.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) have a higher risk than the general population of developing premature cardiovascular disease; the reasons for this are complex. Two recent randomized controlled trials in peritoneal dialysis patients have demonstrated that targeting patients to higher dialysis clearance values is not associated with a reduction in mortality. It is known that patients on peritoneal dialysis are more likely to be volume expanded, develop left ventricular hypertrophy, and have inadequate blood pressure relative to patients on hemodialysis. As a result there has been increased attention on the role of fluid management in reducing the risk of developing congestive heart failure and other adverse cardiovascular events in peritoneal dialysis patients.

Extracellular fluid volume and total body water can be accurately assessed with multi-frequency bioimpedance analysis (BIA). Estimation of volume expansion by measuring the natriuretic peptide N-BNP produced by cardiac tissue in response to ventricular wall stretch can also be used.

The purpose of this study is to determine whether volume status, as measured by BIA and N-BNP levels, correlates with clinical volume assessment, cardiovascular outcomes, peritoneal membrane transport properties and markers of inflammation such as serum albumin and C-reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* 18 years of age or older,
* with end stage renal disease on peritoneal dialysis for a minimum of 3 months

Exclusion Criteria:

* Peritonitis in previous 3 months;
* history of bilateral lower limb amputation;
* inability to provide informed consent;
* presence of a pacemaker or defibrillator;
* anticipated death or transplant within 6 months of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peritoneal dialysis clinic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Brimble, MD, Principal Investigator — McMaster University; Peter Margetts, MD, PhD, Study Director — McMaster University; David N Churchill, MD, MSc, Study Director — McMaster University; Azim S Gangji, MD, Study Director — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Gangji AS, Brimble KS, Margetts PJ. Association between markers of inflammation, fibrosis and hypervolemia in peritoneal dialysis patients. Blood Purif. 2009;28(4):354-8. doi: 10.1159/000232937. Epub 2009 Sep 1. PMID 19729905
- [Result] Gangji AS, Helal BA, Churchill DN, Brimble KS, Margetts PJ. Association between N-terminal propeptide B-type natriuretic peptide and markers of hypervolemia. Perit Dial Int. 2008 May-Jun;28(3):308-11. No abstract available. PMID 18474925